CLINICAL TRIAL: NCT01751490
Title: Does Surgery Followed by Physiotherapy Improve Short and Long Term Outcomes for Patients With Atraumatic Shoulder Instability Compared With Physiotherapy Alone?
Brief Title: Effectiveness of Surgery for Atraumatic Shoulder Instability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Royal National Orthopaedic Hospital NHS Trust (Other)
Collaborators: University of Sydney (Other)
Responsible Party: Principal Investigator, Iva Hauptmannova, Sponsor representative, Royal National Orthopaedic Hospital NHS Trust
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 12.024
Record Dates: First submitted 2012-12-05; First posted 2012-12-18 (Estimated); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Atraumatic Shoulder Instability
Keywords: shoulder; instability; atraumatic
MeSH Terms: interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- physiotherapy alone (Active Comparator): patients undergoing physiotherapy only
  Interventions: Other: physiotherapy; Procedure: shoulder stabilisation surgery
- surgery and physiotherpay (Active Comparator): patients receiving surgical treatment followed by physiotherapy
  Interventions: Other: physiotherapy; Procedure: shoulder stabilisation surgery

INTERVENTIONS:
Other: physiotherapy — physiotherapy
Procedure: shoulder stabilisation surgery — arthroscopic stabilisation surgery
  Other Names: arthroscopic stabilisation surgery

SUMMARY:
We will conduct a randomised clinical trial with the primary aim of determining whether surgical intervention followed by physiotherapy rehabilitation improves pain and disability outcomes more than physiotherapy rehabilitation alone in patients suffering from atraumatic shoulder instability associated with bony/capsulolabral damage. The results of this study will have direct and immediate impact on clinical decision making by establishing definitively if patients presenting with joint damage associated with atraumatic shoulder instability should be referred for surgery before commencing physiotherapy rehabilitation. The results of this study may also result in significant cost savings to the National Health Service if surgical intervention for atraumatic shoulder instability does not result in greater improvement than physiotherapy alone.

DETAILED DESCRIPTION:
A two-arm, patient, physiotherapist and assessor-blinded, randomised controlled clinical trial will be conducted. 140 patients will be randomly allocated into one of 2 groups: a stabilisation surgery group and a control group. Primary outcomes (pain and disability) and secondary outcomes (participant-reported improvement and incidence of shoulder dislocations) will be evaluated at baseline and 6, 12 and 24 months after randomisation. Additional secondary outcomes of shoulder rotation range of motion and strength will be evaluated 6 months after randomisation.

ELIGIBILITY:
Inclusion Criteria:

* feelings of insecurity (apprehension) at their shoulder joint
* provocation of apprehension with drawer and apprehension tests
* evidence labral/capsular injury in the shoulder joint

Exclusion Criteria:

* a history of a high collision shoulder injury precipitating apprehension symptoms
* evidence of bony injury around glenoid rim/and or humeral head
* a pristine joint i.e. no evidence of any structural injury to the joint, capsule or labrum.
* a rotator cuff tear
* neural damage affecting the upper limb
* previous shoulder surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-02; Primary Completion 2022-12 (Actual); Study Completion 2022-12 (Actual)

PRIMARY OUTCOMES:
Change in pain and functional impairment, measured using the Western Ontario Shoulder Instability Index. | over 24 months
  Looking at time points of baseline, 6 months, 12 months and 24 months

SECONDARY OUTCOMES:
Global perceived effect assessing participant-perceived improvement | over 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Anju Jaggi, BSc, Principal Investigator — Royal National Orthopaedic Hospital NHS Trust; Susan Alexander, MD, Principal Investigator — Royal National Orthopaedic Hospital NHS Trust & UCL; Karen Ginn, BSc, PhD, Principal Investigator — University of Sydney; Andrew Symonds, BSc, MSc, Principal Investigator — Royal National Orthopaedic Hospital NHS Trust; Suzie Cro, BSc, Principal Investigator — Royal National Orthopaedic Hospital NHS Trust
Locations (1):
- Royal National Orthopaedic Hospital NHS Trust, Stanmore, Middlesex, United Kingdom

REFERENCES:
- [Derived] Jaggi A, Herbert RD, Alexander S, Majed A, Butt D, Higgs D, Rudge W, Ginn KA. Arthroscopic capsular shift surgery in patients with atraumatic shoulder joint instability: a randomised, placebo-controlled trial. Br J Sports Med. 2023 Dec;57(23):1484-1489. doi: 10.1136/bjsports-2022-106596. Epub 2023 Jun 12. PMID 37308285
- [Derived] Jaggi A, Alexander S, Herbert R, Funk L, Ginn KA. Does surgery followed by physiotherapy improve short and long term outcome for patients with atraumatic shoulder instability compared with physiotherapy alone? - protocol for a randomized controlled clinical trial. BMC Musculoskelet Disord. 2014 Dec 17;15:439. doi: 10.1186/1471-2474-15-439. PMID 25515666
- See also: Royal National Orthopaedics Hospital (RNOH) main website — http://www.rnoh.nhs.uk/